CLINICAL TRIAL: NCT02716220
Title: BIOTRONIKS - Acute Performance Of a Drug Eluting Absorbable Metal Scaffold (DREAMS 2G) in Patients With de Novo Lesions in NatiVE Coronary Arteries: BIOSOLVE-III
Brief Title: Pre-market Study of the DREAMS 2G Drug Eluting Absorbable Metal Scaffold (BIOSOLVE-III)
Acronym: BIOSOLVE-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1502
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis
Keywords: DREAMS 2G; Scaffold; Drug Eluting Absorbable Metal Scaffold; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 'Percutaneous Coronary Intervention' /Scaffold Implantation (Experimental): PCI for enrolled subjects: implantation of the DREAMS 2G Drug-Eluting Coronary Scaffold System
  Interventions: Device: Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — Implanttaion fo the DREAMS 2G Scaffold

SUMMARY:
BIOSOLVE-III Study is a pre-market, prospective, multi-center trial to assess the acute clinical performance of the DREAMS 2G Drug-Eluting Coronary Scaffold in de novo coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years and < 80 years of age
2. Written subject informed consent available prior to PCI
3. Subjects with stable or unstable angina pectoris or documented silent ischemia
4. Subject eligible for PCI
5. Subject acceptable candidate for coronary artery bypass surgery
6. Subjects with a maximum of two single lesions in two separate coronary arteries which have to be de novo lesions.
7. Reference vessel diameter between 2.7-3.8 mm by visual estimation, depending on the scaffold size used.
8. Target lesion length by visual estimation, assisted by QCA: < 21 mm, depending on the scaffold size used.
9. Target lesion stenosis by visual estimation, assisted by QCA > 50% - < 100%
10. Eligible for Dual Anti Platelet Therapy (DAPT)

Exclusion Criteria:

1. Pregnant or breast-feeding females or females who intend to become pregnant during the time of the study
2. Evidence of myocardial infarction within 72 hours prior to index procedure
3. Subjects with a ≥2 fold CK level or in absence of CK a ≥3 fold CKMB level above the upper range limit within 24 hours prior to the procedure
4. Left main coronary artery disease
5. Three-vessel coronary artery disease at time of procedure
6. Thrombus in target vessel
7. Subject is currently participating in another study with an investigational device or an investigational drug and has not reached the primary endpoint yet
8. Planned interventional treatment of any non-target vessel within 30 days post procedure
9. Subjects on dialysis
10. Planned intervention of the target vessel after the index procedure
11. Ostial target lesion (within 5.0 mm of vessel origin)
12. Target lesion involves a side branch >2.0 mm in diameter
13. Documented left ventricular ejection fraction (LVEF) ≤ 30%
14. Heavily calcified lesion
15. Target lesion is located in or supplied by an arterial or venous bypass graft
16. The target lesion requires treatment with a device other than the pre-dilatation balloon prior to scaffold placement (including but not limited to directional coronary atherectomy, excimer laser, rotational atherectomy, etc.)
17. Unsuccessful pre-dilatation, defined as minimal lumen diameter smaller than the respective crossing profile of DREAMS 2G and angiographic complications (e.g. distal embolization, side branch closure, extensive dissections that can't be covered by a single scaffold), by visual estimation
18. Known allergies to: Acetylsalicylic Acid (ASA), Heparin, contrast medium, Sirolimus, Everolimus or similar drugs (i.e., ABT 578, Biolimus, Tacrolimus), PLLA, Silicon Carbide Magnesium, Yttrium, Neodymium, Zirconium, Gadolinium, Dysprosium, Tantalum
19. Impaired renal function (serum creatinine > 2.5 mg/dl or 221mmol/l) determined within 72 hours prior to intervention
20. Subject is receiving oral or intravenous immuno-suppressive therapy ( inhaled steroids are not excluded) or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus)
21. Proximal or distal to the target lesion located stenosis that might require future revascularization or impede run off detected during diagnostic angiography
22. Life expectancy less than 1 year, or other co-morbidities (e.g. Sepsis, Apoplexy or TIA within 6 months prior to the study procedure) (Co-morbidities definitions will be left to the discretion of the Study Investigators)
23. Planned surgery or dental surgical procedure within 6 months after index procedure
24. Subject with tortuous vessel that may impair scaffold placement in the region of obstruction or proximal to the lesion
25. In the investigators opinion subjects will not be able to comply with the follow-up Requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Acute performance of the DREAMS 2G | During the hospital stay to a maximum of 7 days post study Procedure
  Acute performance of the DREAMS 2G assessed by procedure success. Procedure success is defined as: Procedure Success is defined as achievement of a final diameter stenosis of <30% by QCA (using any percutaneous method) without the occurrence of death, Q-wave or non-Q-wave MI, or repeat revascularization of the target lesion during the hospital stay

SECONDARY OUTCOMES:
Target Lesion Failure (TLF) | 1, 6 12, 24 and 36 months post procedure
  TLF defined as a composite of Cardiac Death, Target Vessel Q-wave or non-Q wave Myocardial Infarction (MI)**, Coronary Artery Bypass Grafting (CABG), clinically driven Target Lesion Revascularization (TLR)
Scaffold thrombosis rate | 1, 6 12, 24 and 36 months post procedure
Binary in-scaffold and in-segment restenosis rate | 12-months
% in-scaffold and in-segment diameter stenosis | 12-months
In-segment late lumen loss | 12-months
In-scaffold late lumen loss | 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haude, MD, Principal Investigator — Städtische Kliniken Neuss
Locations (8):
- Interventional Cardiology Middelheim Hospital (ZNA Middelheim), Antwerp, Belgium
- Germany (5):
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Vivantes Klinikum Friederichshain,, Berlin
  - Amper Kliniken AG, Dachau
  - Städtische Kliniken Neuss, Neuss
  - Universitätsmedizin Rostock, Rostock
- Thoraxcenter, Erasmus Medical Center, Rotterdam, Netherlands
- Universitätsklinik Inselspitalspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No